CLINICAL TRIAL: NCT02918370
Title: Aripiprazole for Bipolar Disorder and Alcohol Use Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Sherwood Brown, MD, PhD, Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 102015-062
Record Dates: First submitted 2016-09-27; First posted 2016-09-28 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Bipolar Disorder; Alcoholism; Alcohol Abuse
Keywords: Alcohol Use Disorder; Bipolar Disorder; Mood; Alcohol Craving; Aripiprazole; Schizoaffective Disorder
MeSH Terms: conditions — Bipolar Disorder; Alcoholism; Psychotic Disorders | interventions — Aripiprazole; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aripiprazole (Experimental): Aripiprazole will be given to the participant beginning at 2 mg per day(QD) then titrating up to 5 mg QD at week 1, 10 mg QD at week 2, 15 mg QD at week 3 until the end of the preliminary phase. If the participant qualifies for the extension phase, then they will be titrated up again at week 12 to 30 mg QD.
  Interventions: Drug: Aripiprazole
- Placebo (Placebo Comparator): Matching placebo will be given to the participant beginning at 2mg QD then titrating up to 5 mg QD at week 1, 10 mg QD at week 2, 15 mg QD at week 3 until the end of the preliminary phase. If the participant qualifies for the extension phase, then they will be titrated up again at week 12 to 30 mg QD.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole is an atypical antipsychotic drug that is used to treat mental/mood disorders. It works to restore the balance of neurotransmitters.
  Other Names: Abilify
  Arms: Aripiprazole
Drug: Placebo — Inactive ingredient matching the active comparators in appearance.
  Other Names: Sugar Pill
  Arms: Placebo

SUMMARY:
The investigators will conduct a 12-week, randomized, double-blind, parallel-group, placebo-controlled study of aripiprazole in 132 persons with Alcohol Use Disorder (AUD) and bipolar I or II disorder, currently depressed or mixed phase. Primary Aim will be to assess change in alcohol use by the Timeline Followback (TLFB) method. Secondary Aim will include change in alcohol craving using the Penn Alcohol Craving Scale (PACS). Changes in psychiatric symptoms (mania/hypomania and depression) and predictors of response will be assessed. Participants with ≥ 1 drinking day at week 12 will be enrolled in a 4-week extension phase with an upward titration to 30 mg/day for those in the active treatment group. The placebo group will remain on placebo.

Subjects will be discontinued from the study if any of the following conditions occurs: change in diagnosis to other than bipolar I or II disorder and AUD, development of active suicidal or homicidal ideation with plan and intent, worsening in mood symptoms, that in the opinion of the investigators requires discontinuation, pregnancy, development of severe or life-threatening medical condition, involuntary psychiatric hospitalization or incarceration, significant alcohol withdrawal (e.g. delirium tremens) based on clinical judgment (increases in Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar) scores will initiate a careful clinical assessment of possible worsening of withdrawal symptoms), or cocaine or amphetamine-positive urine drug screen during the study.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient men and women age 18-65 years old with bipolar I, II, Not Otherwise Specified (NOS) disorder, or Schizoaffective Bipolar Type
* If diagnosed with Bipolar I, Bipolar NOS w/history of mania or Schizoaffective Disorder Bipolar Type, current mood stabilizer therapy (lithium, valproic acid, lamotrigine, gabapentin) with stable dose for > 28 days prior to randomization.
* Baseline Barrett Impulsiveness Scale-11 Score of > 62 (above average impulsivity)
* Systolic BP > 100 and < 165 and Diastolic BP > 60 and < 105 with no evidence of orthostatic hypotension
* Current Diagnosis of Alcohol Use Disorder with at least moderate severity
* Alcohol use of an average of 15 drinks per 7 days in the past 28 days prior to intake for men, and an average of 8 drinks per 7 day period in the past 28 days prior to intake for women
* Current mood stabilizer therapy with stable dose for > 28 days
* Fluent in English or Spanish

Exclusion Criteria:

* Baseline Hamilton Rating Scale for Depression (HRSD) or Young Mania Rating Scale (YMRS) scores > 35
* Mood disorders other than bipolar I, II, NOS or schizoaffective disorder bipolar type (e.g. cyclothymic disorders, schizophrenia, schizoaffective disorder depressive type, or unipolar depression based on the SCID), other disorders, e.g. anxiety disorders, will be allowed.
* Current diagnosis of amphetamine or cocaine use disorder or a cocaine or amphetamine positive baseline urine sample.
* Evidence of clinically significant alcohol withdrawal symptoms
* Current treatment with an atypical antipsychotic
* Current treatment with naltrexone, acamprosate, disulfiram, or topiramate in the last 28 days
* Prior treatment with Aripiprazole within the last year or lifetime history of intolerable side effects to Aripiprazole
* Vulnerable populations (e.g. pregnant, nursing, cognitively impaired, incarcerated.)
* Evidence of clinically significant alcohol withdrawal symptoms defined as a CIWA-Ar score of ≥ 10.
* High risk for suicide
* Aspartate Amino Transferase (AST) or Alanine Amino Transferase (ALT) > 3 times upper limit of normal
* Current use of Cytochrome P450 3A4 inducing medication (e.g. carbamazepine, rifabutin, rifampin, ritonavir).
* Use of other substances (besides cocaine/amphetamine) is allowed if the use disorder is no greater than moderate severity and alcohol is the self-identified substance of choice.
* History of neuroleptic malignant syndrome or tardive dyskinesia.

More specific inclusion and exclusion criteria will be discussed with participant at baseline assessment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aripiprazole | Placebo
Started | 36 | 39
Completed | 34 | 30
Not Completed | 2 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Placebo | Total
Number analyzed (Participants) | 36 | 39 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.71 (9.35) | 43.58 (12.25) | 43.65 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 19 | 35
  Male | 20 | 20 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 27 | 28 | 55
  Unknown or Not Reported | 4 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 20 | 34
  White | 20 | 15 | 35
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
TLFB (Drinks per Drinking Day) [Mean (Standard Deviation); unit: standard drinks per drinking day] | 8.42 (5.12) | 10.02 (7.94) | 9.25 (6.74)
HRSD [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale is an observer-rated measure of depressive symptomatology. The individual item scores range from 0-4, 0-3 or 0-2 depending on the question. The higher the score represents greater depressive symptom severity. The possible range of scores is 0-52.
  units on a scale | 13.62 (7.40) | 14.19 (7.56) | 13.82 (7.43)
IDS-SR [Mean (Standard Deviation); unit: units on a scale] — The Inventory of Depressive Symptoms Self Report (IDS-SR) is a 30-item self-report scale of depressive symptoms. Th scores on each item range from 0-3. Higher scores indicate greater depressive symptom severity. The possible range of scores is 0-84.
  units on a scale | 26.03 (15.79) | 30.62 (15.42) | 28.42 (15.66)
YMRS [Mean (Standard Deviation); unit: units on a scale] — The Young Mania Rating Scale (YMRS) is an 11-item, observer-rated measure of manic symptoms. There are four items that are graded on a 0 to 8 scale (irritability, speech, thought content, and disruptive/aggressive behavior), while the remaining seven items are graded on a 0 to 4 scale. These four items are given twice the weight of the others to compensate for poor cooperation from severely ill patients. There are well described anchor points for each grade of severity. The higher score represents a higher level of mania. The possible range of scores is 0-60.
  units on a scale | 8.92 (6.80) | 10.33 (6.96) | 9.85 (7.34)
CIWA-Ar [Mean (Standard Deviation); unit: units on a scale] — The Clinical Institute of Withdrawal Assessment of Alcohol (CIWA-Ar) scale is a 10-item, clinician-rated scale of alcohol withdrawal symptoms. Each item scores range from 0-7. Higher scores indicate greater withdrawal symptom severity. The possible range of scores is 0-67.
  units on a scale | 2.50 (2.67) | 3.05 (3.60) | 2.79 (3.18)
PACS [Mean (Standard Deviation); unit: units on a scale] — The Penn Alcohol Craving Scale (PACS) is a 5-item questionnaire that measures an individual's craving to drink alcohol in the past week. Each item scores range from 0-6. Higher scores indicate greater craving. The possible range of scores is 0-30.
  units on a scale | 19.50 (6.31) | 17.79 (7.53) | 18.60 (6.98)
BIS-11 [Mean (Standard Deviation); unit: units on a scale] — The Barratt Impulsiveness Scale (BIS-11) is a 30 question self-report measure of impulsiveness. It is rated on a four-point Likert scale of 1 = Rarely/Never to 4 = Almost Always/Always. The total scores can range from 30 to 120. Higher scores reflect higher levels of impulsiveness. The possible range of scores is 30-120.
  units on a scale | 79.09 (13.41) | 78.10 (13.34) | 78.56 (13.29)

OUTCOME MEASURES:

1. Primary Outcome: Timeline Follow Back (TLFB)
Description: The Timeline Followback (TLFB) is used to assess recent alcohol use (and if present, other substance use). The calculation is based on the change between baseline and week 12.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: drinks per drinking day
Arm/Group | Aripiprazole | Placebo
Number analyzed (Participants) | 36 | 39
drinks per drinking day | -0.82 (5.86) | -0.71 (4.23)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Aripiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/36 | 2/39
Other Adverse Events (participants affected / at risk) | 13/36 | 5/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=36) | Placebo (N=39)
increased glucose (Metabolism and nutrition disorders) | 0 | 1 — A participant receiving a placebo was hospitalized with high glucose levels. The diagnosis was that pre-diabetes may have progressed to diabetes. Follow-up for further assessment was arranged after discharge.
Flare up of multiple sclerosis (Nervous system disorders) | 0 | 1 — Participant receiving placebo had a flare up of multiple sclerosis requiring hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aripiprazole (N=36) | Placebo (N=39)
Restlessness/Fidgeting (General disorders) | 11 | 2
Increased urinary frequency or difficulty (Renal and urinary disorders) | 2 | 3
Dry mouth (General disorders) | 6 | 1
Headache (Nervous system disorders) | 3 | 3
Nausea or vomiting (Gastrointestinal disorders) | 13 | 4
erectile dysfunction or decreased libido (General disorders) | 0 | 3
increased appetite or weight gain (General disorders) | 4 | 5
Somnolence (General disorders) | 9 | 2
Insomnia (General disorders) | 2 | 3
diarrhea (Gastrointestinal disorders) | 0 | 2
fatigue (General disorders) | 2 | 1
dyspepsia (Gastrointestinal disorders) | 4 | 0
constipation (Gastrointestinal disorders) | 3 | 1
tremors (Nervous system disorders) | 1 | 2
dizziness or lightheadedness (Nervous system disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-19): https://cdn.clinicaltrials.gov/large-docs/70/NCT02918370/Prot_SAP_000.pdf